CLINICAL TRIAL: NCT01630772
Title: Influence of a Physical Therapy Protocol in Maternal and Fetal Hemodynamics in Pregnant Women With Preeclampsia
Brief Title: Physical Therapy in Pregnant Women With Preeclampsia
Acronym: FPE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Tawana Vicente Bertagnolli, physiotherapist graduate student in biology of reproduction, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 6500; 65002010 (Other: Approval of the ethics committee)
Record Dates: First submitted 2012-06-25; First posted 2012-06-28 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Preeclampsia
Keywords: women with preeclampsia; physical therapy; maternal-fetal hemodynamics; perinatal outcomes
MeSH Terms: conditions — Pre-Eclampsia | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Physical therapy — Physical therapy in women with preeclampsia during the hospitalization
  Other Names: Physicotherapy; Hemodinamic
Other: No physical therapy — Comparison of maternal and fetal hemodynamics in women with preeclampsia who underwent physical therapy and who did not have physical therapy
  Other Names: Physiotherapy; Hemodinamic

SUMMARY:
The aim of this study is to evaluate the influence that has a physical therapy protocol in maternal and fetal hemodynamics in relation to blood pressure, maternal and fetal responses and perinatal outcomes.

DETAILED DESCRIPTION:
The hypertensive disorders in pregnancy affecting 5-8% of pregnant women worldwide, contributing significantly to maternal and fetal complications. Various forms of hypertensive disorders occurring during pregnancy, including preeclampsia and chronic hypertension with superimposed preeclampsia. These two disorders present with high blood pressure and proteinuria, and often lead to the hospitalization of pregnant women.

The objective is to evaluate the effectiveness of a physical therapy protocol used in pregnant women with preeclampsia on blood pressure, maternal-fetal outcomes and perinatal outcomes.

Participants in the study pregnant women with preeclampsia and hypertension with superimposed pre-eclampsia, hospitalized, with no significant complications that may impair the normal course of pregnancy. All pregnant women are monitored through laboratory and clinical data and the fetus monitored by tests that assessed their vitality, in addition, pregnant women in the intervention group performed the proposed physiotherapeutic the study protocol.

ELIGIBILITY:
Inclusion Criteria:

Participed of The study, high-risk pregnant women with gestational age between 24 and 38 weeks, hospitalized with a diagnosis of preeclampsia or chronic hypertension with superimposed preeclampsia, with no other maternal diseases and absence of fetal diseases by diagnostic ultrasound examinations and fetal well.

Exclusion Criteria:

* Pregnant women who became symptomatic (blurred vision, epigastric pain, headache) secondary to the hypertensive process;
* 24-hour proteinuria above 2 g
* Laboratory abnormalities (thrombocytopenia, alteration of renal function, elevated liver enzymes, elevated bilirubin);
* Request the patient to leave the project.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-01 (Estimated); Study Completion 2013-02 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital Clinics, University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil